CLINICAL TRIAL: NCT00433979
Title: Predictors of Antiretroviral Pharmacokinetics in HIV-infected Women With Virologic Suppression on Combination Antiretroviral Therapy
Brief Title: Study of Pharmacokinetics in HIV-infected Women
Status: Completed | Type: Observational
Sponsor: Women's College Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Mona Loutfy, Women's College Research Institute
Other Study IDs: HHP-79215
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: HIV Infections
Keywords: Anti-HIV agents; Physiological Effects of Drugs; ARV-associated Adverse Events; HAART; Pharmacokinetics; Protease Inhibitors; Non-nucleoside Reverse Transcriptase Inhibitors; Women
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn before and after antiretroviral drugs are taken for visits 1-3.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: antiretroviral treatment — These antiretroviral drugs are a part of the participant's current drug regimen.

SUMMARY:
Women represent an increasing proportion of HIV cases globally and in Canada, yet are underrepresented in clinic trials. It is therefore critical to conduct this study on antiretroviral (ARV) pharmacokinetics (PK) in women to obtain additional information on ARV drug levels in women and their relation to adverse events (AEs).

The hypothesis for this study is three-fold:

1. that the mean drug levels (Cmin and Cmax) of ARVs will be significantly higher in our female population as compared to the mean drug levels in the historical HIV population (which is primarily men)
2. that ARV drug levels, particularly Cmin, are associated with body weight in women
3. that higher ARV drug levels, particularly Cmax, are associated with higher frequency and severity of AEs.

The objectives of this study are as follows:

Primary objectives:

1. To demonstrate that levels of Protease Inhibitors (PIs) and Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs) are significantly higher in our female population as compared to the mean drug levels in the historical general population (which is primarily men).
2. To determine the association between PI and NNRTI minimum concentration (Cmin) and body weight in our female population.

Secondary objectives

1. To determine the association between maximum concentration (Cmax) and the frequency and severity of AEs as measured by the proportion of patients with grade 2 or higher laboratory or clinical AEs and the Symptom Index Score in women.
2. To determine the association between ARV drug levels and age, race, height, body mass index, adherence, hormonal levels and therapy, menstruation history, duration of HIV infection, duration on ARV therapy, baseline viral load, baseline CD4 count, present CD4 count, hepatitis B or C infection, class of ARVs, presence of ritonavir and other medications.

DETAILED DESCRIPTION:
Predictors of antiretroviral pharmacokinetics in HIV-infected women with virologic suppression on combination antiretroviral therapy

Background

Women in Canada constitute the fastest growing population groups at risk for infection with HIV and AIDS. Women now represent approximately 40% of all AIDS cases worldwide and approximately 20% of cases in Canada. Although the AIDS epidemic has been ongoing for more than 20 years, surprisingly little is known about the differential efficacy and toxicity of various antiretroviral (ARV) drugs in women as compared to men. This gap in knowledge is a result of the initial exclusion of and continued underrepresentation of women in ARV clinical trials. Many studies suggest that HIV-infected women taking ARV treatment (ART) have more adverse events (AEs) than men, especially in relationship to systemic symptoms like diarrhea, as well as organ toxicity, including hepatotoxicity, lactic acidosis, peripheral neuropathy and, notably, lipodystrophy. Currently, the occurrence and management of AEs is the most important issue in the treatment of HIV. Understanding the reasons for the differences of AEs in HIV-infected women is critical and has yet to be evaluated within a large cohort. It is unknown whether these differences relate to hormonal influences, drug metabolism, adherence, fat distribution, body size or other factors. Some small studies have found that drug levels (e.g. Cmin, Cmax, AUC) are higher in women and are associated with increased toxicity. Ultimately, we plan to conduct a randomized clinical trial (RCT) to assess the utility of therapeutic drug monitoring (TDM) and ARV drug dose adjustment on the frequency of AEs in women. Prior to conducting this RCT, it is critical to conduct this study on ARV pharmacokinetics (PK) in women to obtain additional information on ARV drug levels in women and their relation to AEs.

Hypothesis

The hypothesis for this study is three-fold:

1. that the mean drug levels (Cmin and Cmax) of ARVs will be significantly higher in our female population as compared to the mean drug levels in the historical HIV population (which is primarily men)
2. that ARV drug levels, particularly Cmin, are associated with body weight in women
3. that higher ARV drug levels, particularly Cmax, are associated with higher frequency and severity of AEs.

Patient population

Eighty HIV-infected women from 8 Canadian sites who have been on their first combination ART regimen containing either a PI or an NNRTI (since these are the ARV agents eligible for PK analysis) for at least three months and who have evidence of full virologic suppression (HIV RNA VL less than 50 copies/mL) on at least two occasions at least one month apart.

Objectives Primary objectives

1. To demonstrate that the Cmin and Cmax of PIs and NNRTIs are significantly higher in our female population as compared to the mean drug levels in the historical general population (which is primarily men).
2. To determine the association between PI and NNRTI Cmin and body weight in our female population.

Secondary objectives

1. To determine the association between Cmax and the frequency and severity of AEs as measured by the proportion of patients with grade 2 or higher laboratory or clinical AEs and the Symptom index score in women.
2. To determine the association between ARV drug levels and age, race, height, body mass index, adherence, hormonal levels and therapy, menstruation history, duration of HIV infection, duration on ARV therapy, baseline VL, baseline CD4 count, present CD4 count, hepatitis B or C infection, class of ARVs, presence of ritonavir and other medications.

Study design

The study will be a cross-sectional study with ARV drug levels (Cmin and Cmax) measured weekly for three weeks Three samples will be taken from each subject to reduce variability due to both technologic and biologic sources. Data will be collected on demographic characteristics, clinical disease and ARV history and on clinical toxicities at the first visit. Blood work will be carried out on the first visit to assess for laboratory toxicity and hormonal levels.

Data analysis

Drug levels will be summarized with the mean of the 3 values for Cmin and Cmax for each woman for their PI or NNRTI and compared to the mean values of the general HIV population. Cmin and Cmax will be classified into high and low levels with a high level defined as less than or equal to 1.5 X arithmetic population mean for each drug. Characteristics of patients with high drug levels will be compared to those of patients with low drug levels. Univariate and multivariate logistic regression models will be used to identify independent associations of patient characteristics with high drug levels. The proportions of patients with AEs and the median number of AEs per patient will be compared between patients with high Cmax and patients with low Cmax.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be HIV infected
* Patient must be 18 years old or older
* Patient must be a biologic woman
* Patient must be taking her first combination ARV regimen that includes a PI or an NNRTI for the past three months with no changes in any agent of the combination in that period (first combination ARV regimen is defined as a regimen started when the patient was ARV-naïve; however switches are allowed as long as the switches are not for virologic failure)
* Patient must be taking either a PI or an NNRTI but not both
* If taking a PI, patient must be taking only one PI excluding low dose ritonavir used as boosting
* Patient must have a viral load < 50 copies/mL on two occasions at least 1 month apart including a value within three months before the baseline visit
* Patient has to have signed and dated a full informed consent

Exclusion Criteria:

* Patient who would have difficulty participating in a trial due to non-adherence or substance abuse
* Patient who is pregnant or breast-feeding
* Patient with a malignancy receiving systemic chemotherapy
* Patient with end stage organ disease
* Patient with other significant non-HIV underlying disease that might impinge upon disease progression or death
* Patient who is not taking standard dosing of a PI or NNRTI as listed in Appendix G

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will consist of 80 HIV-infected women (who are on their first cART regimen containing either a PI or an NNRTI for at least three months and who have evidence of full virologic suppression (HIV RNA VL < 50 copies/mL) on at least two occasions at least one month apart. The first cART regimen can include ARV switches as long as these switches are not due to virologic failure. The patient population is being limited to women who have full virologic suppression to avoid inclusion of women with difficulty with drug adherence.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mona R Loutfy, MD FRCPC MPH, Principal Investigator — Women's College Hospital
Locations (15):
- Canada (15):
  - Children and Women's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Downtown Infectious Diseases Clinic, Vancouver, British Columbia
  - Capital District Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences - McMaster University, Hamilton, Ontario
  - University of Ottawa Health Services, Ottawa, Ontario
  - Ottawa Health Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Canadian Immunodeficiency Research Collaborative, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Windsor Regional Hospital HIV Care Program, Windsor, Ontario
  - Centre de recherche du Centre hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Montreal Chest Institute, Montreal, Quebec
  - Chuq/Chul, Québec, Quebec

REFERENCES:
- [Derived] Loutfy MR, Walmsley SL, Klein MB, Raboud J, Tseng AL, Blitz SL, Pick N, Conway B, Angel JB, Rachlis AR, Gough K, Cohen J, Haase D, Burdge D, Smaill FM, de Pokomandy A, Loemba H, Trottier S, la Porte CJ. Factors affecting antiretroviral pharmacokinetics in HIV-infected women with virologic suppression on combination antiretroviral therapy: a cross-sectional study. BMC Infect Dis. 2013 Jun 3;13:256. doi: 10.1186/1471-2334-13-256. PMID 23732043